CLINICAL TRIAL: NCT06769360
Title: A Pragmatic Pilot Trial Evaluating Inspiratory Pressure Adjustment Based on Pressure Muscle Index in Patients Undergoing Pressure Support Ventilation
Brief Title: A Pilot Trial of Pressure Muscle Index-Targeted PSV Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-206-02
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Critical Care; Acute Hypoxic Respiratory Failure; Ventilator Lung
Keywords: pressure support ventilation; pressure muscle index; inspiratory effort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PMI-targeted group (Experimental): Will be treated by standard of care for patients undergoing mechanical ventilation (e.g., protective PSV settings, protocolized weaning, etc.) + pressure support is adjusted according to PMI between 0 and 2 cmH2O during PSV.
  Interventions: Procedure: PMI-targeted PSV setting
- VT/RR-targeted group (Active Comparator): Will be treated by standard of care for patients undergoing mechanical ventilation (e.g., protective PSV settings, protocolized weaning, etc.).
  Interventions: Procedure: VT/RR-targeted PSV setting

INTERVENTIONS:
Procedure: PMI-targeted PSV setting — The pressure support is adjusted according to PMI between 0 and 2 cmH2O. After application of PSV mode in mechanically ventilated patients, the initial PS level was first set based on respiratory rate (RR) <35 beats/min and 6-8 ml/Kg tidal volume (Vt) per predict body weight (PBW), and then modified according to PMI at a frequency of twice a day (morning and afternoon bedside rounds)# 1) Perform three end- inspiratory occlusions, with at least 1 minute between each measurement, and calculate the mean PMI. 2) Determine whether the PMI is within the target range (0≤PMI≤2cmH2O). 3) If the PMI is not within the target range, adjust the PS level up or down by 1-3 cmH2O and balance for 3-5 minutes. 4) Repeat the above steps until PMI reaches the target. 5) Additional: During PS adjustment, if Vt≤4ml/Kg, respiratory acidosis, respiratory distress, Vt≥8ml/Kg, respiratory alkalosis occurs, return to the safe PS level before adjustment and optimize other treatments.
  Arms: PMI-targeted group
Procedure: VT/RR-targeted PSV setting — Standard of care: the pressure support is adjusted to obtain a VT between 6 and 8 ml/kg PBW and RR between 20 and 35 breaths/min.
  Arms: VT/RR-targeted group

SUMMARY:
Pressure support ventilation (PSV) is one of the most frequently used ventilator modes in the intensive care unit (ICU). The successful implementation of PSV depends on matching the patient's inspiratory effort with the ventilator support. In clinical practice, the pressure support level is usually set and adjusted according to tidal volume (VT) and respiratory rate (RR). However, these parameters may not fully represent the patient's effort. Previous studies have shown that pressure muscle index (PMI), which is measured as the difference between the peak and plateau airway pressure during an end-inspiratory airway occlusion, could reliably determine the low and high inspiratory effort during PSV.

However, the comparative effectiveness of these two pressure support level setting strategies remains uncertain. Our aim is to explore clinical and implementation factors relevant to a future definitive randomized controlled trial to evaluate PMI - and VT/RR - pressure support level setting strategies. The Inspiratory effort-targeted pressure support ventilation pragmatic pilot trial will test clinician adherence and to explore clinical outcomes.

Two centers are included in a pragmatic sequential cluster crossover pilot trial. We enrolled all eligible adults with acute respiratory failure requiring mechanical ventilation admitted to ICU. The pressure support level setting strategy was assigned according to the epoch. The first trial epoch will be assigned to VTRR - pressure support level setting strategy for 4 weeks. The washout week between the two epochs will be 4 weeks. Then sequentially, it will be crossed over to PMI - pressure support level setting strategy for 4 weeks.

* In the VT/RR-targeted group, the pressure support is adjusted to obtain a VT between 6 and 8 ml/kg PBW and RR between 20 and 35 breaths/min until day 28 or death or performance of spontaneous breathing trial (SBT).
* In the PMI-targeted group, the pressure support is adjusted according to PMI between 0 and 2 cmH2O until day 28 or death or performance of SBT.

We will also survey clinicians to understand potential facilitators and barriers to conducting a definitive randomized trial.

DETAILED DESCRIPTION:
Steering committee (chief investigators): Feng-Xue Zhu, Li Weng, Jian-Xin Zhou

Aim.

Our aim is to explore clinical and implementation factors relevant to a future definitive randomized controlled trial to evaluate PMI - and VT/RR - pressure support level setting strategies. The Inspiratory effort-targeted pressure support ventilation pragmatic pilot trial will test clinician adherence and to explore clinical outcomes.

Study design and Work plan.

Two centers are included in a pragmatic sequential cluster crossover pilot trial. The pressure support level setting strategy will be assigned according to the epoch. The first trial epoch will be assigned to VTRR - pressure support level setting strategy for 4 weeks, because that is the current standard practice in ICU prior to study initiation. The washout week between the two epochs will be 4 weeks. Then sequentially, it will be crossed over to PMI - pressure support level setting strategy for 4 weeks. Before each epoch, a one-week comprehensive training program will be conducted for all staff in the participating ICUs.

Patients

Mechanically ventilated patients admitted to the ICU with acute hypoxic respiratory failure (AHRF) will be consecutively screened daily at 08:00-10:00 morning rounds. Patients undergoing PSV are eligible for inclusion. The patients will be enrolled only once during the same hospitalization. Written informed consent will be obtained from the patient or their legal representative.

Study Procedures

In both PMI-targeted and VT/RR-targeted groups, standard clinical care for mechanical ventilation is followed according to local routine practice, which is formatted based on international clinical guidelines, except for pressure support adjustment during PSV.

General standard of care for mechanical ventilation

Analgesia is routinely used in mechanically ventilated patients with continuous infusion of fentanyl or remifentanil. Sedation with midazolam, propofol, or dexmedetomidine is used when the patient exhibits agitation and a light sedation level is maintained on RASS of -2 to +1 or Riker's SAS of 3 to 4.

In patients with AHRF, mechanical ventilation is usually initiated on protective control ventilation, such as volume or pressure control mode, with VT 6-8 ml/kg predicted body weight (PBW), RR to control arterial partial pressure of carbon dioxide (PaCO2) and pH, and FiO2 and PEEP to maintain pulse arterial oxygen saturation (SpO2) between 90% and 95%.

Transition of control modes to PSV

During the morning rounds, the responsible ICU physicians check the ventilator mode for each patient. The ventilator mode is recommended to transit from controlled modes to PSV if all the following criteria are met:

1. The patient is able to trigger ventilator breaths;
2. PaO2/FiO2 above 100 mmHg;
3. PEEP below 15 cmH2O;
4. Stable hemodynamic status (none or stable doses of vasopressors);
5. No sedation or light sedation ([RASS] of -2 to +1 or [SAS] of 3 to 4).

PSV setting strategy

In both the PMI-targeted and VT/RR-targeted groups, the same principle PSV settings are followed except for the adjustment of pressure support level:

1. The inspiratory trigger sensitivity is set as 1-2 L/min for the flow-trigger or 1.5-3 cmH2O for the pressure-trigger;
2. Inspiration-to-expiration cycle-off is set as 25% of the peak inspiratory flow. Responsible physicians can adjust this parameter in case of suspected cycle-off patient-ventilator asynchrony;
3. FiO2 and PEEP are set to maintain SpO2 between 90% and 95%. Specifically, if SpO2 is lower than 90%, PEEP and then FiO2 will be increased by 2 cmH2O and 0.1, respectively; whereas if SpO2 is higher than 95%, FiO2 and then PEEP will be decreased by 0.1 and 2 cmH2O, respectively.

In the VT/RR-targeted group, the pressure support is adjusted to obtain a VT between 6 and 8 ml/kg PBW, RR between 20 and 35 breaths/min, and no signs of respiratory distress, such as prominent use of the accessory respiratory muscles, nose flaring, retractions, etc.

In the PMI-targeted group, the pressure support is adjusted according to the PMI between 0 and 2 cmH2O. During PSV, after an end-inspiratory airway occlusion, Paw will reach a plateau. PMI can be measured on the ventilator screen as plateau Paw minus peak Paw by using a sliding marking line when the screen frozen function is initiated. According to our previous studies, a PMI value of 0 to 2 cmH2O will be used as the target for pressure support adjustment. This PMI range represents a well-accepted normal inspiratory effort.

During the study period in the two groups, pressure support adjustment will be performed at least twice daily.

Rescue backup of controlled ventilation

In both groups, PSV can be switched to protective controlled modes when predefined criteria are met, which include at least one of the following conditions:

1. Pressure support level above 20 cmH2O;
2. PEEP above 15 cmH2O;
3. pH < 7.30;
4. PaO2/FiO2 ≤ 100 mmHg;
5. Strong inspiratory effort which cannot be controlled by sedation;
6. Unstable hemodynamic status (systolic blood pressure below 90 mmHg with vasopressors or systolic blood pressure above 180 mmHg);
7. Active cardiac ischemia;
8. Unconsciousness (RASS < -3 or SAS < 2);
9. Dangerous agitation that cannot be controlled by sedation (RASS > +2 or SAS > 6).

Data will be documented in patients whose mechanical ventilation is switched to controlled modes. The patients will be reassessed at least every 12 hours and transited back to PSV as soon as possible according to the abovementioned criteria. The patients will be visited daily until 28 days after randomization. Data will be documented and reported for those patients whose controlled ventilation is not transited back to PSV during the follow-up.

Weaning and extubation

The weaning and extubation process follows clinical guidelines recommended by the American Thoracic Society and the American College of Chest Physicians.

The attending physicians assess readiness to initiate the weaning process during daily morning rounds. If all the following aspects are satisfied, an SBT will be performed:

1. Improvement of the cause of intubation and mechanical ventilation;
2. Hemodynamic stability when the dose of norepinephrine is less than 0.1 μg/kg/min or equivalent and lasts for 6 hours at stable or reduced doses;
3. No agitation or coma;
4. SpO2 higher than 90% with FiO2 less than 0.4 and PEEP less than 5 cmH2O.

SBT is conducted by respiratory therapists using the low-level PSV with pressure support of 5 cmH2O and PEEP of 5 cmH2O. The SBT will last at least 30 min, and criteria for failure of SBT include:

1. RR of greater than 35 breaths/min for more than 5 min;
2. SpO2 of less than 90%;
3. Elevated PaCO2 and/or pH of less than 7.3;
4. Heart rate (HR) of greater than 140 beats/min or a sustained change in HR of more than 20%;
5. Systolic blood pressure greater than 180 mmHg or less than 90 mmHg;
6. Signs of cardiac ischemia indicated by dynamic ST changes on ICU monitor or electrocardiogram;
7. Abrupt unconsciousness with RASS below -3 or SAS below 2;
8. Signs of anxiety, agitation, or diaphoresis. Patients with a failure SBT will be mechanically ventilated with PSV following settings and adjustments according to the original grouping.

Extubation will be performed in endotracheal intubated patients who pass the SBT, and mechanical ventilation will be discontinued in patients with tracheostomy. PSV will be restored to maintain the grouping in patients with reintubation or reapplication of mechanical ventilation via tracheostomy within seven days. The decision to reintubate and restore mechanical ventilation will be at the discretion of the ICU physician team according to the local standard of care. The duration of mechanical ventilation will be added to the total duration.

Data Collection

An electronic case report form (eCRF) is designed and available online via Electronic Data Capture System (Yiduoyun medical health corporation, suzhou, china).

Data collected at the study entry

At baseline, demographics, comorbidities, diagnosis for ICU admission, recent medical history, reasons for mechanical ventilation, duration of ventilation before enrolment, conditions of gas exchange, and mechanical ventilation settings will be documented, as will the Acute Physiological and Chronic Health Evaluation II (APACHE II) score at the ICU admission.

Data collection during daily visits

All patients will be visited daily between 08:00 and 12:00 until successful weaning or separation of mechanical ventilation, death, hospital discharge, or until 28 days after randomization. Successful weaning or separation of mechanical ventilation is defined as extubation without reintubation or death within the next seven days, whether post-extubation noninvasive ventilation is used or not, or ICU discharge without invasive mechanical ventilation within seven days, whichever comes first.

Data collected include:

1. Gas exchange: SpO2 and arterial blood gas analysis;
2. Hemodynamics: blood pressure, HR, vasoactive agents, and cumulative fluid balance during the last day;
3. Analgesia and sedation: RASS or SAS score, visual analog scale or critical care pain observation tool, the use of analgesics and sedatives;
4. Sequential Organ Failure Assessment (SOFA) score;
5. Switch to controlled ventilation: whether switching to controlled mode during the last 24 hours, reasons, and settings;
6. PSV: pressure support level, PEEP, FiO2, VT, and RR;
7. Respiratory drive: the negative airway pressure generated during the first 100 ms against an end-expiratory airway occlusion (airway occlusion pressure, P0.1) (29);
8. SBT: whether performing an SBT during the last 24 hours, methods, and results;
9. Extubation or discontinuation of mechanical ventilation: whether performed during the last 24 hours;
10. Re-intubation or restoration of mechanical ventilation: whether performed during the last 24 hours and reasons;
11. Tracheostomy: whether performed during the last 24 hours;
12. Self-extubation: whether occurring during the last 24 hours;
13. 28-day follow-up: duration of mechanical ventilation, length of stay in the ICU and hospital, and death.

After the study, a questionnaire survey will be conducted involving all staff members in the participating ICUs. The survey mainly includes Likert scales to assess the PMI - pressure support level setting strategy acceptability and also assessed feasibility of conducting a full RCT. Additionally, we also have open-ended questions to understand the difficulties in implementation and ways to improve compliance.

ELIGIBILITY:
Inclusion Criteria:

1. PSV initiated during the last 24 hours, whether transition from controlled modes or primary initiation;
2. Mechanical ventilation expected to be required for at least 24-48 hours by responsible physicians;
3. The partial pressure of oxygen in arterial blood (PaO2)/inspired oxygen fraction (FiO2) ≤ 300 mmHg (measuring at clinical FiO2 and positive end-expiratory pressure [PEEP]);
4. No sedation or stable sedation with Richmond Agitation Sedation Scale (RASS) of -2 to +1 or Riker's Sedation-Agitation Scale (SAS) of 3 to 4.

Exclusion Criteria:

1. Age younger than 18 years old;
2. Initiation of PSV before ICU admission;
3. Duration of mechanical ventilation longer than 7 days before enrollment;
4. History of neuromuscular diseases;
5. Clinical suspicion of increased intracranial pressure;
6. Presentation with pneumothorax and/or bronchopleural fistula;
7. Extracorporeal support;
8. Moribund conditions;
9. Refusal by the ICU physicians or the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PMI target pressure support level setting strategy | 1 year
  Defined as 75% of the test points in which PMI can reach 0-2 cmH2O.

SECONDARY OUTCOMES:
Feasibility of VT/RR target pressure support level setting strategy | 1 year
  Defined as 75% of the test points in which VT can reach 6-8 ml/kg PBW and RR can reach 20-35 breaths/min.
Ventilator-free days (VFDs) | 1 year
  ventilator-free days (VFDs) at day 28 after enrollment. This analysis will be performed comparing the 2 study groups.
Duration of mechanical ventilation before enrollment | 1 year
  Defined as the mechanical ventilation time before enrollment. This analysis will be performed comparing the 2 study groups.
Total duration of mechanical ventilation | 1 year
  Defined as the time intervals from intubation to successful weaning. For patients with re-intubation or restoration of mechanical ventilation via tracheostomy within 72 hours after extubation and discontinuation of ventilation, the thereafter duration will be added. This analysis will be performed comparing the 2 study groups.
The time before the first SBT | 1 year
  Defined as the time interval from intubation and mechanical ventilation to the first SBT attempt.This analysis will be performed comparing the 2 study groups.
Weaning time | 1 year
  defined as the time from the first SBT attempt to successful discontinuation of mechanical ventilation. This analysis will be performed comparing the 2 study groups.
Frequency of prolonged weaning | 1 year
  Defined following WIND classification. This analysis will be performed comparing the 2 study groups.
Frequency of self-extubation, re-intubation, tracheotomy, and mechanical ventilation longer than 21 days | 1 year
  Compare the incidence of these adverse events in the 2 study groups.
Length of stay in the ICU and hospital | 1 year
  This analysis will be performed comparing the 2 study groups.
ICU mortality, hospital mortality, and 28-day mortality | 1 year
  This analysis will be performed comparing the 2 study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No